CLINICAL TRIAL: NCT05983887
Title: The Effect of Therapeutic Climbing on Muscle Strength, Tone and Balance in Hemiplegic Children: a Preliminary Single-blind Randomised Controlled Trial
Brief Title: The Effect of Therapeutic Climbing on Muscle Strength, Tone and Balance in Hemiplegic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pavlos Kitixis (Other)
Responsible Party: Sponsor-Investigator, Pavlos Kitixis, Principal Investigator, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: climb_in_hem
Record Dates: First submitted 2023-07-30; First posted 2023-08-09 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2024-05

CONDITIONS: Hemiplegia and Hemiparesis
Keywords: therapeutic climbing; hemiplegia; children; muscle strength; balance
MeSH Terms: conditions — Hemiplegia; Paresis

STUDY DESIGN:
Intervention Model Description: Single-blind Randomised Controlled Trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The participants in this group continue their conventional intervention protocol without using the climbing instructions.
- Climbing Group (Experimental): The participants in this group continue their conventional intervention protocol plus an in-door climbing intervention protocol.
  Interventions: Other: Therapeutic Climbing

INTERVENTIONS:
Other: Therapeutic Climbing — The protocol consists of using an in-door climbing wall as an complementary therapeutic intervention model.
  Arms: Climbing Group

SUMMARY:
The goal of this randomised controlled trial is to learn about the effect of therapeutic climbing in hemiplegic children. The main questions it aims to answer are:

Does climbing affect muscle strength and tone? What is its connection between normative data drawn from healthy children? How can it affect balance?

Participants (children) will be asked to complete an series of movements used in sports climbing, such as inside-flag, back-flag and horizontal traverse, while hanging on an in-door climbing wall.

ELIGIBILITY:
Inclusion Criteria:

* Children from 4 to 16 years old
* Children with Hemiplegia
* Evaluated as Level 1 on GMFCS

Exclusion Criteria:

* Botulinum toxin injection in last 6 months
* Surgery in the last 1 year (myofascial lengthening etc.)
* Children with poor cognitive skills (not following instructions etc.)

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | 8 weeks (pre-post evaluation)
  Measured using Kinvent K-PUSH Dynamometer and Jamar Hydraulic Hand Dynamometer ; Unit of Measure: Peak Force in Kilograms (higher scores - better outcome)
Balance | 8 weeks (pre-post evaluation)
  Measured using the Timed Up & Go Test ; Unit of Measure: seconds of completion (higher scores - worse outcome)
Muscle Tone | 8 weeks (pre-post evaluation)
  Evaluated using the Modified Ashworth Scale ; Unit of Measure: Scoring Options (0-4) // (higher scores - worse outcome)

SECONDARY OUTCOMES:
Normative Strength Data Comparison | 8 weeks (pre-post evaluation)
  Comparison of normative values of the Jamar Hydraulic Hand Dynamometer of Healthy and Hemiplegic Children ; Unit of Measure: Difference of Peak Force in Kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Besios, PhD, Study Chair — University of Thessaly
Locations (1):
- Department of Physiotherapy, Lamia, Phthiotis, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buechter RB, Fechtelpeter D. Climbing for preventing and treating health problems: a systematic review of randomized controlled trials. Ger Med Sci. 2011;9:Doc19. doi: 10.3205/000142. Epub 2011 Aug 9. PMID 21863133
- See also: The effect of therapeutic climbing on gross motor function in hemiplegic cerebral palsy. A pilot single-case experimental design study (SCED) — https://www.researchgate.net/publication/325380027_The_effect_of_therapeutic_climbing_on_gross_motor_function_in_hemiplegic_cerebral_palsy_A_pilot_single-case_experimental_design_study_SCED